CLINICAL TRIAL: NCT03328715
Title: iOCT in Patients With Diabetic Macular Edema Scheduled for Phakoemulsification - a Pilot Study
Brief Title: iOCT for Patients With Diabetic Macular Edema
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vienna Institute for Research in Ocular Surgery (Other)
Responsible Party: Principal Investigator, Prim. Prof. Dr. Oliver Findl, MBA, Prim, Prof.,, Vienna Institute for Research in Ocular Surgery
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: DMÖ-iOCT
Record Dates: First submitted 2017-10-29; First posted 2017-11-01 (Actual); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: Diabetic Macular Edema

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Active Comparator): only patients with diabetic macular edema will be recruited in that arm, stand-alone OCT and intraoperative OCT will be performed before and after surgery
  Interventions: Device: intraoperative OCT; Device: stand-alone OCT
- controll group (Sham Comparator): only patients without diabetic macular edema will be recruited in that arm, stand-alone OCT and intraoperative OCT will be performed before and after surgery
  Interventions: Device: intraoperative OCT; Device: stand-alone OCT

INTERVENTIONS:
Device: intraoperative OCT — before and after surgery intraoperative OCT is performed
Device: stand-alone OCT — before and after surgery stand-alone OCT is performed

SUMMARY:
Patients will be examined before and after surgery with a stand-alone OCT and intraoperative microscope integrated OCT

DETAILED DESCRIPTION:
48 patients with and 48 patients without diabetic macular edema will be recruited for the study. Macular thickness measured with a stand-alone OCT and an intraoperative OCT will be assessed before and after phakoemulsification with intraocular lens Implantation.

ELIGIBILITY:
Inclusion Criteria:

* Cataract with the indication for surgery (visual symptoms) for both groups (study and control group)
* Diabetic macula edema - for the study group
* Age 21 and older
* written informed consent prior to surgery

Exclusion Criteria:

* Any relevant corneal disease
* In case of pregnancy (pregnancy test will be taken preoperatively in women of reproductive age)

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2016-12-01 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
macular thickness | 2 hours
  macular thickness is measured with the central subfield thickness function

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Findl, MD, Prof, Principal Investigator — Vienna Institute for Research in Ocular Surgery
Locations (1):
- Vienna Institute for Research in Ocular Surgery (VIROS), Hanusch Hospital Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No